CLINICAL TRIAL: NCT04636151
Title: E-Manage: A Brief mHelath Intervention for University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Evan M. Kleiman, Ph.D., Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2020002347
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Distress, Emotional; Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual Treatment (Experimental): Participants will have up to three individual sessions with a study therapist. One or more treatment modules will be presented in each session.
  Interventions: Behavioral: Ecological momentary intervention
- Group Treatment (Experimental): Participants will have up to three group sessions with a study therapist. One or more treatment modules will be presented in each session.
  Interventions: Behavioral: Ecological momentary intervention
- Workshops (Experimental): Participants will have one workshop with a study therapist. All three treatment modules will be presented in one session.
  Interventions: Behavioral: Ecological momentary intervention

INTERVENTIONS:
Behavioral: Ecological momentary intervention — Content of this intervention is based on pre-established transdiagnostic protocols for addressing the negative emotion associated with suicidal thoughts and behaviors.

SUMMARY:
This study is a two-part transdiagnostic psychological intervention aimed to help people respond to negative emotion and emotional distress in more adaptive ways using a technology called "ecological momentary intervention" (or EMI) that delivers intervention content using a smartphone app. Participants in this study will be Rutgers students recruited through-or currently affiliated with - Counseling, Alcohol and Other Drug Assistance Program & Psychiatric Services (CAPS) at Rutgers. Participants will first attend either one-on-one or group telehealth therapy sessions/workshops, where they will learn the therapeutic skills that are part of the study. Then, they will complete up to 8 weeks of smartphone monitoring that involves assessments and opportunities to practice the skills learned in therapy.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older
* Matriculated at Rutgers during Fall of 2020 (on campus and/or remote)
* Currently residing in US
* Willingness to follow study requirements, as evidenced by an ability to provide written informed consent and read, understand, and complete the study procedures
* iOS and Android smartphone compatible with MetricWire. Nearly all phones since 2014 are compatible

Exclusion Criteria

* Non-English speaking
* Unable to understand or provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in momentary levels of self-reported distress | 8 week study period
  Assessed via smartphone assessments

SECONDARY OUTCOMES:
Change in momentary levels of suicidal thinking | 8 week study period
  Assessed via smartphone assessments

CONTACTS AND LOCATIONS:
Overall Officials: Evan Kleiman, Ph.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Counseling, Alcohol and Other Drug Assistance Program & Psychiatric Services (CAPS), Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the informed consent and de-identified data.
Supporting Information: ICF
Time Frame: We will share the informed consent after the final participant has enrolled. We will share de-identified data one year after the study is finished.

DOCUMENTS (1):
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT04636151/ICF_000.pdf